CLINICAL TRIAL: NCT03234426
Title: Effectiveness of Perturbations Exercises in Improving Balance, Function and Mobility in Stroke Patients.
Acronym: perturbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahatma Gandhi Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nawaj Pathan, M.P.Th.PG student, Mahatma Gandhi Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MGM ECRHS 2014/160
Record Dates: First submitted 2014-12-10; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): manual perturbations were given in forward, Backward,right and left sideways, 10 perturbations were given,6 days in week,in fallowing positions- sitting,kneeling, standing positions
  Interventions: Other: Perturbation; Other: Conventional Physiotherapy Treatment
- Control group (Placebo Comparator): Conventional Physiotherapy were given 6 days in a week, for 30 mins for 4 weeks, includes stretching, strengthening of contralateral limbs
  Interventions: Other: Perturbation; Other: Conventional Physiotherapy Treatment

INTERVENTIONS:
Other: Perturbation — Manual perturbations were given at waist region,over the Shoulders. in following positions- sitting, kneeling, standing positions,10 perturbations were given in forward,backward,both right and left side, 6 days in a week all precautionary measures taken for the patient's safety
  Other Names: Manual Perturbation
Other: Conventional Physiotherapy Treatment — Conventional Physiotherapy treatment were given to participants included in this group for 30 mins daily for 4 weeks
  Other Names: control Group

SUMMARY:
Following stroke, patients loses functions of the motor, sensory and higher brain cognitive faculties to various degrees which lead to diminished balance. It has been documented that hemiplegic or hemiparetic stroke patients presented with more posture sway, asymmetric weight distribution, impaired weight-shifting ability and decreased stability capability. There are many balance exercises and strategies; to improve balance in elderly age group population, to prevent fall prevention. But we have very few evidences of giving manual perturbation balance training in stroke patients to improve speed, balance and function. Therefore this study is taken up to examine whether the manual perturbation balance training is more effective in improving speed, balance and function in stroke patients.

DETAILED DESCRIPTION:
There are many more studies done for elderly populations, normal individuals for improving balance by giving perturbation based balance training.All perturbation exercises are given by either mechanical or by self reaching tasks in forward,backward,and in both sideways. There are very studies ;who attempted perturbation based balance training to improve balance in elderly population but not for stroke patients for their Speed, Balance and Function.The manual perturbation exercise can be an promising intervention in the future for various conditions

ELIGIBILITY:
Inclusion Criteria:

1. First ever stroke
2. Age ranges between 40-70
3. Both genders were included
4. Ambulatory patients with or without ambulatory aids
5. Occurrence of stroke at within 0-3 months i.e.-sub acute
6. Able to follow command
7. Mini mental scale examinations not less than 24

Exclusion Criteria:

1. Patients who has severe limitations in passive range of motion at lower extremities
2. Patients with impaired sensory, proprioceptor, cognitive and perceptual ability
3. Patient who has contracture
4. Orthopedic or any other neurological disorder which impair balance

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 4 weeks
  patients ability of balance were assessed

SECONDARY OUTCOMES:
Functional Independence Scale | 4 weeks
  ability of Functional independent level for Activity Of Daily Living were assessed

OTHER OUTCOMES:
Timed Up and Go Test | 4 weeks
  patient's speed for performing Activity Of Daily Living were assessed by this test

CONTACTS AND LOCATIONS:
Overall Officials: Nawaj Pathan, PG student, Principal Investigator — MGM School Of Physiotherapy,Aurangabad,Maharashtra, India
Locations (1):
- MGM school Of Physiotherapy, Aurangabad, Maharashtra, India